CLINICAL TRIAL: NCT07081815
Title: A Single Center Clinical Trial Investigating the Safety and Efficacy of JOCOAT(TM) APN-3003 Liquid Adhesion Barrier Device for Knee Anterior Cruciate Ligament Reconstruction Surgery
Brief Title: JOCOAT Safety and Tolerability Clinical Trial GLAD-04
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ARC Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ARCMD-GLAD-04
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Surgical Adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: All patients in this study will receive the investigational treatment. Safety and clinical outcomes from this study will be compared with historical controls from enrolled study site patients from NCT03935750.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JOCOAT(TM) APN-3003 (Experimental): Intra-articular injection
  Interventions: Device: JOCOAT(TM) APN-3003

INTERVENTIONS:
Device: JOCOAT(TM) APN-3003 — 10 mL of JOCOAT(TM) APN-3003 is applied at the end of surgery

SUMMARY:
This study will assess the safety and efficacy of a new liquid anti-adhesion device, JOCOAT(TM) APN-3003 in patients undergoing knee anterior cruciate ligament reconstruction (ACLR) surgery.

This is a single-center, prospective study. Safety and clinical outcomes will be compared with historical controls from enrolled study site patients from NCT03935750 (STABILITY 2) which has evaluated outcomes following ACL rupture in young athletes.

A maximum of 24 patients aged 15-25 years undergoing primary anatomic ACLR with quadriceps tendon (QT) graft following a standardized surgical treatment algorithm will be enrolled. All patients will receive JOCOAT(TM) APN-3003 at the end of their surgery.

ELIGIBILITY:
Pre-operative Inclusion Criteria:

* Understand and be able to follow the requirements of the protocol including personally signing and dating an REB approved Informed Consent Form prior to undergoing any protocol related procedures
* Subjects aged 15 to 25 years with an ACL-deficient knee undergoing primary ACLR
* Subjects with skeletal maturity (i.e. closed epiphyseal growth plates on standard knee radiographs)
* At least two of the following factors that are associated with a high risk of graft failure:

  1. participate in a competitive pivoting sport (defined as sports that include cutting and pivoting activities such as basketball, American football, soccer, lacrosse, volleyball, tennis/squash, handball, downhill skiing etc);
  2. have a pivot shift of grade 2 or greater;
  3. have generalized ligamentous laxity (Beighton score of >= 4) and/or genu recurvatum > 10 degrees
* Biological females have a negative pregnancy test within 4 days of initial surgery
* Is willing, able and likely to fully comply with clinical trial procedures and restrictions including follow-ups

Pre-operative Exclusion Criteria:

* Simultaneous bilateral ACLR
* Previous ACLR on either knee
* Less than one year from contralateral knee or contralateral/ipsilateral hip/ankle surgery
* Prior arthrotomy in the study knee
* Active infection anywhere or previous infection in the study knee
* History of peri-articular fracture in study knee
* > 3 degrees of asymmetric varus or valgus
* The patient has debilitating knee pain that would preclude the use of QT tissue as a graft
* The patient has a significant quad tendonitis that would preclude the use of QT tissue as a graft
* Known or suspected allergy to brown seaweed, seaweed-based materials such as fucoidan, food allergies and/or presence of any allergy related dietary restrictions unless deemed by the investigator as "Not Clinically Significant"
* Known or suspected allergy to fucose, galactose, sulfur, sulfate, sulfite, or any sugar-based polymer or polysaccharides containing these
* Known hypersensitivity to sodium lactate or sulfur-containing compounds
* Any other severe allergic conditions or previous reactions (e.g., anaphylactic reactions, angioedema)
* Severe metabolic acidosis or alkalosis
* Have insulin dependent diabetes, severe diabetes and/or poorly controlled diabetes mellitus
* Any general medical or surgical condition that would preclude a standard knee ACLR
* Inflammatory arthropathy
* Breast feeding
* Have a medical condition that, in the opinion of the investigator would interfere with the evaluation of the safety or efficacy of the investigational product
* Have received any investigational products that, in the opinion of the investigator, would interfere with the evaluation of the safety or efficacy of the investigational product
* Have clinically relevant hemochromatosis, hepatic, renal, autoimmune, lymphatic, hematological or coagulation disorders
* Family history of blood or coagulation disorders
* History of heparin-induced thrombocytopenia (HIT) or known sensitivity to heparin-like products

Intra-operative Inclusion Criteria:

- Patient undergoes primary anatomic anterior cruciate ligament reconstruction surgery with quadriceps tendon (QT) graft

Intra-operative Exclusion Criteria:

* Pre-existing arthrofibrosis in the knee
* Partial ACL rupture (defined as one bundle ACL tear requiring reconstruction/ augmentation of the torn bundle with no surgery required for the intact bundle) where ACLR is not performed
* Multiple ligament injury (two or more ligaments requiring surgery)
* Symptomatic articular cartilage defect requiring treatment other than debridement
* Articular cartilage lesion that requires any other surgical treatment apart from debridement
* Under anesthetic, this patient has a symmetrical or grade 1 pivot shift AND has a Beighton score <4 AND <10 degrees hyperextension

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety of JOCOAT(TM) APN-3003 as measured by number and severity of adverse device effects and serious adverse device effects | 3 months after surgery
  The number of severe and serious adverse events in treated subjects from this study is compared with the number seen in historical controls

SECONDARY OUTCOMES:
Exploratory efficacy of JOCOAT(TM) APN-3003 as measured by comparing range of motion (ROM) pre-operatively and post-operatively | 3 months after surgery
  Range of motion is measured pre-operative and post-operatively and compared
Patient recovery as measured by Patient Reported Outcome Measures (KOOS) | Up to 12 months after surgery
  Patient reported outcome measure results (Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire) pre-operatively and post-operatively are compared with historical controls
Patient recovery as measured by Patient Reported Outcome Measures (PASS) | Up to 12 months after surgery
  Patient reported outcome measure results (Patient-Acceptable Symptom States (PASS) questionnaire) pre-operatively and post-operatively are compared with historical controls
Patient recovery as measured by Patient Reported Outcome Measures (EQ-5D-5L) | Up to 12 months after surgery
  Patient reported outcome measure results (EQ-5D-5L questionnaire) pre-operatively and post-operatively are compared with historical controls